CLINICAL TRIAL: NCT05015010
Title: Phase II, Open-label, Single-arm, Multicenter Study to Assess the Activity and Safety of ALectinib as NEO-adjuvant Therapy in Patients With Anaplastic Lymphoma Kinase-positive (ALK+) Locally Advanced Stage III Non-Small Cell Lung Cancer (NSCLC): ALNEO Trial
Brief Title: Alectinib in Neo-adjuvant Treatment of Stage III NSCLC
Acronym: ALNEO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-01-2020
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: ALK-positive; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alectinib (Experimental): The treatment will be administrated as neoadjuvant 8 weeks before surgery. After surgical intervention the treatment will be administered up to 96 weeks. Treatment will be discontinued in case of unacceptable toxicity or disease progression.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — 600 mg p.o. (four 150 mg capsules) twice daily with food (within 30 minutes after a meal, in the morning and evening).

SUMMARY:
Stage III NSCLC is a heterogeneous group of tumors with a wide spectrum of clinical presentations. Across this wide spectrum of heterogeneity, there is no single deﬁnitive therapeutic approach and the definition of the most effective treatment approach needs a multidisciplinary approach. In this trial we want to test in ALK positive stage III locally advanced NSCLC patients, the efficacy of Alectinib to induce tumor shrinkage when administered before surgery and to reduce the possibility of disease recurrence, with a limited risk of toxicity related, in long term administration after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed adenocarcinoma of the lung. Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Documented ALK-positive disease according to an FDA-approved and CE-marked test.
* Locally advanced NSCLC in stage III according to the 8th American Joint Committee on Cancer TNM edition, defined potentially resectable (any T with N2, T4N0-1).
* Documentation that the patient is a candidate for surgical resection of their lung cancer after multidisciplinary discussion.
* Patients must be treatment-naive for NSCLC and eligible to receive treatment with Alectinib.
* Measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria with CT scan.
* Brain magnetic resonance imaging (MRI) or CT scan showing no evidence of metastatic disease.
* Positron emission tomography (PET)-computed tomography (CT) showing radiographic stage III lung cancer (mediastinal staging biopsy is allowed but not required).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1.
* Ability to swallow oral medications.
* Adequate haematological function defined by white blood cell (WBC) count ≥ 2.500/mm3 with absolute neutrophil count (ANC) ≥ 1.500/mm3, platelet count ≥ 100.000/mm3 and haemoglobin ≥ 9 g/dL.
* Adequate hepatic function defined by a total bilirubin ≤ 1.5 x the upper limit of normal (ULN) range (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL), serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 if liver function test elevations are due to liver metastases).
* Adequate renal function defined by a serum creatinine ≤ 1.5 x ULN or an estimated creatinine clearance of ≥ 30 mL/minute for patients with creatinine levels above institutional limits (if using the Cockcroft-Gault formula).
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before trial inclusion date, and otherwise noted in other inclusion/exclusion criteria.
* Female patients with childbearing potential should be using adequate contraceptive measures and should not be breastfeeding during the study and for 90 days following the last dose of Alectinib. They and must have a negative serum pregnancy test within 7 days prior to the first dose of study drug.
* Female patients must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments;
  * Women under 50 years old would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment with LH and FSH levels in the post-menopausal range for the institution;
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception for at least 14 days prior to administration of the first dose of study treatment, during the study, and for 90 days following the last dose of Alectinib.
* Ability to comply with protocol requirements.
* Ability to provide written informed consent. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior treatment with any systemic anti-cancer therapy for locally advanced NSCLC including chemotherapy, biologic therapy, including ALK-TKI, immunotherapy or any investigational drug.
* Non-resectable stage III and stage IV disease with distant metastases (including malignant pleural effusion) identified on PET-CT scan or biopsy.
* Any concurrent and/or active malignancy that has required treatment within 2 years of the first dose of study drug.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol; or known active infection including hepatitis B (HBV), hepatitis C (HCV) and human immunodeficiency virus (HIV); screening for chronic conditions is not required; patients with HBV with negative HBV viral load on appropriate antiviral therapy will be permitted, if able to continue appropriate antiviral therapy throughout treatment period.
* Any severe infection, including COVID-19, within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infections.
* History of organ transplant.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of Alectinib.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc)>470 msec, obtained from 3 electrocardiograms (ECGs)
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250msec, symptomatic bradycardia <45 beats/minute.
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
* Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry.
* History of hypersensitivity to active or inactive excipients of Alectinib or drugs with a similar chemical structure or class to Alectinib. This includes, but is not limited to, patients with galactose intolerance, a congenital lactase deficiency or glucose-galactose malabsorption.
* Administration of strong/potent cytochrome P450 (CYP)3A inhibitors or inducers within 14 days prior to the first dose of study treatment and while on treatment with Alectinib except for oral corticosteroids up to 20 mg of prednisolone equivalent per day.
* Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site).
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | From the treatment start until surgery - 12 weeks period (8 weeks of neoadjuvant therapy; surgery should be done within 2-4 weeks afterwards.
  Percentage of residual viable tumor cells histologically detected in the resected primary tumor and all resected lymph nodes after surgery ≤10%. Evaluation by Blinded Independent Pathology Reviewer (BIPR).

SECONDARY OUTCOMES:
Pathological Complete Response | From the treatment start until surgery - 12 weeks period (8 weeks of neoadjuvant therapy; surgery should be done within 2-4 weeks afterwards.
  The absence of residual viable tumor cells in all surgical specimens (resected primary tumor and all resected lymph nodes) as evaluated by BIPR.
Objective response | Pre-surgical radiological evaluation (after 8 weeks of neoadjuvant therapy start)
  Complete Response (CR) or a Partial Responses (PR) based on the Investigator's assessment and measured according to standard RECIST criteria v1.1
Event-free survival (EFS) | From the trial inclusion date to either the date of disease recurrence/progression or the date of death, monitored up to 3 years after surgery.
  The length of time after the trial inclusion the patient remains free of recurrence/progression or death, whatever the cause.
Disease-free survival (DFS) | From the date of surgical resection to either the date of disease recurrence or the date of death monitored up to 3 years after surgery.
  The length of time after surgical resection the patient remains free of recurrence/progression or death, whatever the cause.
Overall survival (OS) | From the date of trial inclusion to the date of death monitored up to 3 years after surgery.
  The length of time after the trial inclusion the patient remains alive
Adverse Events (AE) | From the date of the trial inclusion until 30 days (90 days in case of AE serious/special interest) after the final dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first
  Untoward medical events occurring after trial inclusion. Adverse Events are defined and graded according to Common Terminology Criteria for Adverse Events [CTCAE] version 5.0.
  Adverse event of special interest are cases of potential drug-induced liver, suspected transmission of an infectious agent by the study treatment, Interstitial Lung Disease.
  Serious adverse events is any AE occurring at any dose that results in death; is life-threatening (i.e., in the opinion of the Investigator, the subject is at immediate risk of death from the AE); requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay); results in persistent or significant disability/incapacity (a substantial disruption of the subject's ability to conduct normal life functions); is a congenital anomaly/birth defect; constitutes an important medical event.
Tissue and cell-free (plasma) biomarkers | From the time of diagnosis up to 3 years after surgery
  Characterization of Anaplastic Lymphoma Kinase fusion partner on DNA extracted from tissue biopsy and on cell-free nucleic acid (cfNA) (both cfDNA and cfRNA) extracted from plasma sample.

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - I.R.S.T., Meldola, Forlì-Cesena
  - UOC Oncologia Medica Ospedale Versilia USL Toscana Nord Ovest, Lido di Camaiore, Lucca
  - A.S.S.T - Monza Ospedale San Gerardo, Monza, Monza Brianza
  - Centro di Riferimento Oncologico (CRO) - IRCCS Aviano, Aviano, Pordenone
  - SSD oncologia polmonare - AOU San Luigi Gonzaga, Orbassano, Torino
  - IRCCS Istittuo Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliero Universitaria Policlinico S.Orsola-Malpighi, Bologna
  - Oncologia Medica - PO Rodolico -AOU "Policlinico - Vittorio Emanuele", Catania
  - SODc Oncologia Medica - Azienda Ospedaliera-Universitaria Careggi, Florence
  - Oncologia Medica 2 - IRCCS AOU Policlinico San Martino - IST, Genova
  - Dipartimento Oncologia e Ematologia - Azienda Ospedaliero-Universitaria di Modena, Modena
  - U.O.C Pneumologia ad Indirizzo Oncologico - Azienda Ospedaliera Dei Colli, Napoli
  - Istituto Oncologico Veneto (IOV), Padua
  - UOC di Oncologia Medica - AOU di Parma, Parma
  - Ospedale S. Maria della Misericordia, Perugia
  - IFO Istituto Regina Elena, Roma
  - UOSD Pneumologia Oncologica- Ospedale San Camillo, Roma
  - Fondazione Policlinico Universitario 'A. Gemelli' IRCCS. Università Cattolica del Sacro Cuore, Roma
  - Humanitas Research Hospital - Medical Oncology, Rozzano
  - Dipartimento di Oncologia Medica - Università di Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Detterbeck FC, Boffa DJ, Kim AW, Tanoue LT. The Eighth Edition Lung Cancer Stage Classification. Chest. 2017 Jan;151(1):193-203. doi: 10.1016/j.chest.2016.10.010. Epub 2016 Oct 22. PMID 27780786
- [Background] Huber RM, De Ruysscher D, Hoffmann H, Reu S, Tufman A. Interdisciplinary multimodality management of stage III nonsmall cell lung cancer. Eur Respir Rev. 2019 Jul 8;28(152):190024. doi: 10.1183/16000617.0024-2019. Print 2019 Jun 30. PMID 31285288
- [Background] Postmus PE, Kerr KM, Oudkerk M, Senan S, Waller DA, Vansteenkiste J, Escriu C, Peters S; ESMO Guidelines Committee. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv1-iv21. doi: 10.1093/annonc/mdx222. No abstract available. PMID 28881918
- [Background] Nicholson AG, Chansky K, Crowley J, Beyruti R, Kubota K, Turrisi A, Eberhardt WE, van Meerbeeck J, Rami-Porta R; Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The International Association for the Study of Lung Cancer Lung Cancer Staging Project: Proposals for the Revision of the Clinical and Pathologic Staging of Small Cell Lung Cancer in the Forthcoming Eighth Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Mar;11(3):300-11. doi: 10.1016/j.jtho.2015.10.008. Epub 2015 Dec 24. PMID 26723244
- [Background] Rocco G, Nason K, Brunelli A, Varela G, Waddell T, Jones DR. Management of stage IIIA (N2) non-small cell lung cancer: A transatlantic perspective. J Thorac Cardiovasc Surg. 2016 May;151(5):1235-8. doi: 10.1016/j.jtcvs.2016.01.035. Epub 2016 Mar 17. No abstract available. PMID 26997100
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Yoon SM, Shaikh T, Hallman M. Therapeutic management options for stage III non-small cell lung cancer. World J Clin Oncol. 2017 Feb 10;8(1):1-20. doi: 10.5306/wjco.v8.i1.1. PMID 28246582
- [Background] Lewis J, Gillaspie EA, Osmundson EC, Horn L. Before or After: Evolving Neoadjuvant Approaches to Locally Advanced Non-Small Cell Lung Cancer. Front Oncol. 2018 Jan 23;8:5. doi: 10.3389/fonc.2018.00005. eCollection 2018. PMID 29410947
- [Background] NSCLC Meta-analysis Collaborative Group. Preoperative chemotherapy for non-small-cell lung cancer: a systematic review and meta-analysis of individual participant data. Lancet. 2014 May 3;383(9928):1561-71. doi: 10.1016/S0140-6736(13)62159-5. Epub 2014 Feb 25. PMID 24576776
- [Background] Situ D, Lin Y. Neoadjuvant strategy for stage IIIA-N2 non-small cell lung cancer: chemoradiation or chemotherapy alone? J Thorac Dis. 2017 Sep;9(9):2746-2748. doi: 10.21037/jtd.2017.08.23. No abstract available. PMID 29221230
- [Background] Muller IB, de Langen AJ, Giovannetti E, Peters GJ. Anaplastic lymphoma kinase inhibition in metastatic non-small cell lung cancer: clinical impact of alectinib. Onco Targets Ther. 2017 Sep 13;10:4535-4541. doi: 10.2147/OTT.S109493. eCollection 2017. PMID 28979145
- [Background] Hida T, Nokihara H, Kondo M, Kim YH, Azuma K, Seto T, Takiguchi Y, Nishio M, Yoshioka H, Imamura F, Hotta K, Watanabe S, Goto K, Satouchi M, Kozuki T, Shukuya T, Nakagawa K, Mitsudomi T, Yamamoto N, Asakawa T, Asabe R, Tanaka T, Tamura T. Alectinib versus crizotinib in patients with ALK-positive non-small-cell lung cancer (J-ALEX): an open-label, randomised phase 3 trial. Lancet. 2017 Jul 1;390(10089):29-39. doi: 10.1016/S0140-6736(17)30565-2. Epub 2017 May 10. PMID 28501140
- [Background] Peters S, Camidge DR, Shaw AT, Gadgeel S, Ahn JS, Kim DW, Ou SI, Perol M, Dziadziuszko R, Rosell R, Zeaiter A, Mitry E, Golding S, Balas B, Noe J, Morcos PN, Mok T; ALEX Trial Investigators. Alectinib versus Crizotinib in Untreated ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Aug 31;377(9):829-838. doi: 10.1056/NEJMoa1704795. Epub 2017 Jun 6. PMID 28586279
- [Background] Sakamoto H, Tsukaguchi T, Hiroshima S, Kodama T, Kobayashi T, Fukami TA, Oikawa N, Tsukuda T, Ishii N, Aoki Y. CH5424802, a selective ALK inhibitor capable of blocking the resistant gatekeeper mutant. Cancer Cell. 2011 May 17;19(5):679-90. doi: 10.1016/j.ccr.2011.04.004. PMID 21575866
- [Background] Vavala T, Novello S. Alectinib in the treatment of ALK-positive non-small cell lung cancer: an update on its properties, efficacy, safety and place in therapy. Ther Adv Med Oncol. 2018 Aug 3;10:1758835918789364. doi: 10.1177/1758835918789364. eCollection 2018. PMID 30090122
- [Background] Lin JJ, Riely GJ, Shaw AT. Targeting ALK: Precision Medicine Takes on Drug Resistance. Cancer Discov. 2017 Feb;7(2):137-155. doi: 10.1158/2159-8290.CD-16-1123. Epub 2017 Jan 25. PMID 28122866
- [Background] Song Z, Wang M, Zhang A. Alectinib: a novel second generation anaplastic lymphoma kinase (ALK) inhibitor for overcoming clinically-acquired resistance. Acta Pharm Sin B. 2015 Jan;5(1):34-7. doi: 10.1016/j.apsb.2014.12.007. Epub 2015 Jan 24. PMID 26579422
- [Background] Kodama T, Hasegawa M, Takanashi K, Sakurai Y, Kondoh O, Sakamoto H. Antitumor activity of the selective ALK inhibitor alectinib in models of intracranial metastases. Cancer Chemother Pharmacol. 2014 Nov;74(5):1023-8. doi: 10.1007/s00280-014-2578-6. Epub 2014 Sep 10. PMID 25205428
- [Background] Seto T, Kiura K, Nishio M, Nakagawa K, Maemondo M, Inoue A, Hida T, Yamamoto N, Yoshioka H, Harada M, Ohe Y, Nogami N, Takeuchi K, Shimada T, Tanaka T, Tamura T. CH5424802 (RO5424802) for patients with ALK-rearranged advanced non-small-cell lung cancer (AF-001JP study): a single-arm, open-label, phase 1-2 study. Lancet Oncol. 2013 Jun;14(7):590-8. doi: 10.1016/S1470-2045(13)70142-6. Epub 2013 Apr 30. PMID 23639470
- [Background] Gadgeel SM, Gandhi L, Riely GJ, Chiappori AA, West HL, Azada MC, Morcos PN, Lee RM, Garcia L, Yu L, Boisserie F, Di Laurenzio L, Golding S, Sato J, Yokoyama S, Tanaka T, Ou SH. Safety and activity of alectinib against systemic disease and brain metastases in patients with crizotinib-resistant ALK-rearranged non-small-cell lung cancer (AF-002JG): results from the dose-finding portion of a phase 1/2 study. Lancet Oncol. 2014 Sep;15(10):1119-28. doi: 10.1016/S1470-2045(14)70362-6. Epub 2014 Aug 18. PMID 25153538
- [Background] Shaw AT, Gandhi L, Gadgeel S, Riely GJ, Cetnar J, West H, Camidge DR, Socinski MA, Chiappori A, Mekhail T, Chao BH, Borghaei H, Gold KA, Zeaiter A, Bordogna W, Balas B, Puig O, Henschel V, Ou SI; study investigators. Alectinib in ALK-positive, crizotinib-resistant, non-small-cell lung cancer: a single-group, multicentre, phase 2 trial. Lancet Oncol. 2016 Feb;17(2):234-242. doi: 10.1016/S1470-2045(15)00488-X. Epub 2015 Dec 19. Erratum In: Lancet Oncol. 2017 Mar;18(3):e134. doi: 10.1016/S1470-2045(17)30077-3. PMID 26708155
- [Background] Ou SH, Ahn JS, De Petris L, Govindan R, Yang JC, Hughes B, Lena H, Moro-Sibilot D, Bearz A, Ramirez SV, Mekhail T, Spira A, Bordogna W, Balas B, Morcos PN, Monnet A, Zeaiter A, Kim DW. Alectinib in Crizotinib-Refractory ALK-Rearranged Non-Small-Cell Lung Cancer: A Phase II Global Study. J Clin Oncol. 2016 Mar 1;34(7):661-8. doi: 10.1200/jco.2015.63.9443. Epub 2015 Nov 23. PMID 26598747
- [Background] Yang JC, Ou SI, De Petris L, Gadgeel S, Gandhi L, Kim DW, Barlesi F, Govindan R, Dingemans AC, Crino L, Lena H, Popat S, Ahn JS, Dansin E, Golding S, Bordogna W, Balas B, Morcos PN, Zeaiter A, Shaw AT. Pooled Systemic Efficacy and Safety Data from the Pivotal Phase II Studies (NP28673 and NP28761) of Alectinib in ALK-positive Non-Small Cell Lung Cancer. J Thorac Oncol. 2017 Oct;12(10):1552-1560. doi: 10.1016/j.jtho.2017.06.070. Epub 2017 Jul 6. PMID 28689043
- [Background] Novello S, Mazieres J, Oh IJ, de Castro J, Migliorino MR, Helland A, Dziadziuszko R, Griesinger F, Kotb A, Zeaiter A, Cardona A, Balas B, Johannsdottir HK, Das-Gupta A, Wolf J. Alectinib versus chemotherapy in crizotinib-pretreated anaplastic lymphoma kinase (ALK)-positive non-small-cell lung cancer: results from the phase III ALUR study. Ann Oncol. 2018 Jun 1;29(6):1409-1416. doi: 10.1093/annonc/mdy121. PMID 29668860
- [Background] Pataer A, Kalhor N, Correa AM, Raso MG, Erasmus JJ, Kim ES, Behrens C, Lee JJ, Roth JA, Stewart DJ, Vaporciyan AA, Wistuba II, Swisher SG; University of Texas M. D. Anderson Lung Cancer Collaborative Research Group. Histopathologic response criteria predict survival of patients with resected lung cancer after neoadjuvant chemotherapy. J Thorac Oncol. 2012 May;7(5):825-32. doi: 10.1097/JTO.0b013e318247504a. PMID 22481232
- [Background] Zhang C, Li SL, Nie Q, Dong S, Shao Y, Yang XN, Wu YL, Yang Y, Zhong WZ. Neoadjuvant Crizotinib in Resectable Locally Advanced Non-Small Cell Lung Cancer with ALK Rearrangement. J Thorac Oncol. 2019 Apr;14(4):726-731. doi: 10.1016/j.jtho.2018.10.161. Epub 2018 Nov 5. PMID 30408570
- See also: Lung Cancer Survival Rates: 5-Year Survival Rates for Lung Cancer — https://www.cancer.org/cancer/lung-cancer/detection-diagnosis-staging/survival-rates.html
- See also: National Comprehensive Cancer Network. Non-small cell lung cancer (Version 3.2020). — https://www.nccn.org/professionals/physician_gls/pdf/nscl.pdf